CLINICAL TRIAL: NCT06121453
Title: P50 Supplement: Improving Medications Adherence Equitably Among Patients With Metastatic Breast Cancer and Cardiovascular Disease
Brief Title: Adherence Intervention in Patients With Metastatic Breast Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Claire Sathe, MD, Assistant Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU9129; P50MD017341 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm: Adherence Intervention (Experimental): Multicomponent Adherence Intervention
  Interventions: Behavioral: Multicomponent Adherence Intervention

INTERVENTIONS:
Behavioral: Multicomponent Adherence Intervention — multi-part intervention to reduce barriers to medication use

SUMMARY:
To evaluate the preliminary efficacy of a multicomponent adherence intervention focused on enhancing digital equity and pharmaco-equity among nonadherent patients with metastatic breast cancer (MBC) and cardiovascular disease (CVD) risk factors on endocrine therapy (ET), CDK4/6 inhibitor (CDK 4/6i), and CVD medications. To assess the acceptability and appropriateness of this intervention in patients with MBC and CVD risk factors through validated measures of implementation outcomes. To gain a deeper understanding of the impact of social determinants of health (SDOH) on medication nonadherence through semi-structured interviews with a subset of study participants.

ELIGIBILITY:
Inclusion Criteria:

* Women or men age >18 years
* Diagnosed with stage IV/metastatic breast cancer prescribed endocrine therapy and a CDK4/6i
* Prescribed at least 1 antihypertensive or statin medication for CVD prevention or treatment
* Self-report of at least some nonadherence ET/CDK4/6i or CVD medication on nonadherence screener or verbally to a treating clinician, or nonadherent to ET, CDK4/6i, and/or CVD medication on pharmacy fill data in the EHR (proportion of days covered over prior 180 days <80%).

Exclusion Criteria:

* Non-English or Non-Spanish speaking
* Not cognitively able to complete study requirements
* Inability to provide informed consent for any other reason (e.g, severe psychiatric illness, active substance use)
* Unavailable for 28 weeks of follow-up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants on multicomponent adherence intervention | at 28 weeks
  To determine the preliminary efficacy of a multicomponent adherence intervention that targets digital and pharmaco-equity among patients with metastatic breast cancer with at least some nonadherence to endocrine therapy, CDK4/6 inhibitor, and/or at least one oral cardiovascular disease (CVD) medication (either blood pressure or statin medication), based on its impact on concurrent adherence to endocrine therapy, CDK4/6 inhibitor, and to CVD medication at 28 weeks (or at time of progression of MBC, if prior to 28-week timepoint), assessed by a combination of self-report using the Voils DOSE Nonadherence measure and pharmacy fill data using pharmacy dispensing records available in the Electronic Health Record (EHR).

SECONDARY OUTCOMES:
Changes in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 at 28 weeks | at 28 weeks
  Healthcare related quality of life (HRQOL), measured by the Patient-Reported Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) measuring health-related quality of life. Raw scores (range 1-5 for each question) are translated into T-scores for each domain (physical function, depression, pain intensity, etc) so that the values follow a normal distribution with a population mean T-score of 50 and a standard deviation of 10. Higher scores can mean better or worse outcomes depending on the domain reported.
  Outcomes Measurement Information System (PROMIS)-29.
Digital Health Literacy Scale | at 28 weeks
  A measure of the basic skills necessary for using digital health services, as assessed by a 3-item questionnaire (questions from the Health Information National Trend Survey (HINTS). Scores range with a higher score indicating better level of literacy.(Health Information National Trend Survey). To score the 3-item digital health care literacy scale, we used a sum score of all the items (range 0-4 for each item, sum score range 0-12) such that higher scores indicated higher digital health care literacy.
Number in using the Voils DOSE Nonadherence measure | at 28 weeks
  Number of and intensity of reasons for nonadherence using the Voils DOSE Nonadherence measure (note: reasons include side-effects and perceived need for medications).
Changes in Medical Adherence Self-Efficacy Scale (MASES) at 28 Weeks | at 28 weeks
  Self-efficacy with medication regimen, as measured by the Medical Adherence Self- Efficacy Scale (MASES-R). The Medication Adherence Self-Efficacy Scale (MASES). Each question from the 12-item measure is score from 1-4, and the total score for this scale is calculated as the average score of all the items, such that the minimal total score is 1 and the maximal total score is 4. Higher scores indicate higher medication adherence self-efficacy.
total number of medications and number of doses per day | at 28 weeks
  Medications and regimen complexity

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No